CLINICAL TRIAL: NCT00005731
Title: Develop and Implement Asthma Controlling Strategies
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4940
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-04

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

STUDY DESIGN:
Observational Model: Natural History

SUMMARY:
To develop and implement asthma-controlling educational strategies for inner city and high risk populations.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is a serious chronic disease affecting about 12 million Americans; about 3 million are children. The study was part of an initiative, "Developing and Implementing at the State and Local Level Educational Strategies and Interventions for Controlling Asthma in Inner City and High Risk Populations", released in February 1993 by the National Asthma Education Program of the Office of Prevention, Education and Control.

DESIGN NARRATIVE:

A computer-assisted multimedia instructional and feedback system, "Asthma Patient/Provider Partnership System" (APPPS), was developed for African American and Hispanic school-age children that was suited for adoption and implementation in clinical and other settings based on the National Asthma Education Program's Expert Panel Guidelines on the Diagnosis and Management of Asthma. A formative evaluation of the educational intervention was conducted. Also, an efficacy study of the intervention in three clinical settings was conducted and the findings of this study were incorporated into the APPPS. Finally, a recommended dissemination strategy was prepared for diffusion of the system to other settings.

ELIGIBILITY:
No eligibility criteria

Min Age: 0 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-09; Study Completion 1997-05

REFERENCES:
- [Background] Bartholomew LK, Gold RS, Parcel GS, Czyzewski DI, Sockrider MM, Fernandez M, Shegog R, Swank P. Watch, Discover, Think, and Act: evaluation of computer-assisted instruction to improve asthma self-management in inner-city children. Patient Educ Couns. 2000 Feb;39(2-3):269-80. doi: 10.1016/s0738-3991(99)00046-4. PMID 11040726
- [Background] Bartholomew LK, Shegog R, Parcel GS, Gold RS, Fernandez M, Czyzewski DI, Sockrider MM, Berlin N. Watch, Discover, Think, and Act: a model for patient education program development. Patient Educ Couns. 2000 Feb;39(2-3):253-68. doi: 10.1016/s0738-3991(99)00045-2. PMID 11040725